CLINICAL TRIAL: NCT01651715
Title: Multicentre, Randomised, Double-blind, Parallel, Placebo-controlled Study Evaluating the Efficacy and Safety of Early Self-Treatment of Viral Upper Respiratory Tract Infections With Homeopathic Oral Antibodies to the TLR3 FYW Peptide (TAO1)
Brief Title: Efficacy and Safety Study of Homeopathic Oral Antibodies to Treat Viral Upper Respiratory Tract Infections
Acronym: ESTUAR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Theranor s.p.r.l (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESTUAR001
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAO1, oral homeopathic antibodies (Experimental): TAO1 is an investigational medicinal product containing homeopathic dilutions (<10-24M) of antibodies purified from the serum of rabbit immunised against a synthetic peptide with an amino acid sequence selected in the human toll-like receptor type 3 sequence (anti-TLR3). It is intended for the treatment of viral Upper Respiratory Tract Infections (URTIs) such as common cold, influenza or influenza-like illnesses.
  Interventions: Drug: TAO1, oral homeopathic antibodies
- Placebo (Placebo Comparator): Same characteristics as investigational medicinal Product except for homeopathic dilutions of oral antibodies to the TLR3 FYW peptide
  Interventions: Drug: TAO1, oral homeopathic antibodies

INTERVENTIONS:
Drug: TAO1, oral homeopathic antibodies — TAO1 comprises a mixture of homeopathic dilutions C12+C30+C200 (drug product is made by impregnation of pre-made tablets).
  The investigational product will be taken for 7 days as follow:
  Day 1: 3 tablets over the first 2 hours of treatment, then 3 tablets over the rest of Day 1.
  Days 2-3: 5 tablets/day (intakes distributed evenly over the daytime). Days 4-7: 3 tablets/day (intakes distributed evenly over the daytime).

SUMMARY:
The purpose of this study is to determine whether early self-treatment with homeopathic dilutions of oral antibodies to a key-protein of the immune system are effective and safe in the treatment of viral upper respiratory tract infections

DETAILED DESCRIPTION:
TAO1 is an investigational medicinal product containing homoeopathic dilutions (<10-24M) of antibodies purified from the serum of rabbit immunised against a synthetic peptide with an amino acid sequence selected in the human toll-like receptor type 3 sequence (anti-TLR3). It is intended for the treatment of viral Upper Respiratory Tract Infections (URTIs) such as common cold, influenza or influenza-like illnesses.

The validity of the TAO1 development approach was addressed in a proof of concept study of efficacy in a non-lethal influenza infection in mice. In this blinded study, TAO1 was given in drinking water for 5 days before and 10 days after viral challenge. The statistical analysis of preclinical data was carried out by using the Mann-Whitney non-parametric test (2-tailed). The clinical disease duration was significantly reduced from 6.0 (5.25 (25th percentile);7.0 (75th percentile)) days to 5.0 (5.0;5.0) days (p=0.00037) as well as the overall disease severity that was lowered from 8.0 (7.0;10.0) points to 6.0 (5.0;7.5) points (p=0.00032).

Given the high homoeopathic dilution, the active substance in the finished product lies beyond sensitivity of existing analytical assays. TAO1 is therefore not amenable to pharmacokinetics studies.

There are currently no data on clinical efficacy of TAO1 in common cold obtained in double-blind placebo-controlled clinical trials. Based on the efficacy in the animal model, the expected magnitude of effect of TAO1 in humans is a reduction of common cold duration by 2-3 days, provided that the treatment is started early after the onset of the symptoms.

Primary objective:

To evaluate the efficacy of TAO1 in reducing the severity of symptoms of common cold in otherwise healthy adults.

Secondary objectives:

To evaluate the efficacy of TAO1 in reducing the duration of common cold. To evaluate the impact of TAO1 on health-related Quality of Life (functional impairment) in patients with common cold.

To evaluate the safety of TAO1.

Experimental design: Double-blind, parallel-group, randomised, multicentre, placebo-controlled study.

Treatment allocation: Balanced allocation between TAO1 and placebo (1:1).

At Visit 1, the medications, questionnaires and diary cards will be dispensed to patients who have signed informed consent. Upon contracting a common cold, they will start the treatment immediately and take contact with the doctor by phone within 36 hours. On Day 2-3 after the onset of disease, they will visit the doctor (Visit 2) to confirm the diagnosis. The doctor will check if questionnaires are filled in correctly. On the 10-14th day (at the latest) after start of treatment, Visit 3 is planned to pick up questionnaires, evaluate safety, disease complications and treatment compliance.

Treatment group: TAO1 tablets (to be dissolved in the mouth, not to be swallowed; should be taken at least 10 minutes apart from meals and/or smoking):

Day 1: 3 tablets to be taken over the first 2 hours of treatment, then 3 tablets over the rest of Day 1,

Days 2-3: 5 tablets/day (intakes distributed evenly over the daytime),

Days 4-7: 3 tablets/day (intakes distributed evenly over the daytime).

Control: Placebo tablets: same dosage regimen as for TAO1.

Concomitant medications: Only oral analgesics/antipyretics, such as paracetamol or ibuprofen, will be allowed in case of fever or headache. Each intake of such medications will be registered in the patient's diary.

Severity and duration of self-reported symptoms evaluated daily by the validated Wisconsin Upper Respiratory Symptom Survey short version (WURSS-21)

Evaluation of safety: adverse events (AEs) and serious adverse events (SAEs) coded using the Medical Dictionary for Regulatory Activities (MedDRA) assessed according to their frequency, severity, outcome and relationship to the study drug.

Data collection: Paper Case Report Form (CRF).

Duration of treatment: 7 days

Duration of study: maximum 10 months.

Number of Investigators: about 35 investigators (General Practitioners).

Type of study: Phase II, self-contained study

Number of patients: 240 (120 treated with TAO1 and 120 treated with placebo)

Sample size justification: A sample size of 115 in each group will have 80% power to detect a difference in mean AUCs of 103 (a difference of 30% between a Placebo AUC mean of 310 and a TAO1 AUC mean of 207) assuming that the common standard deviation is 277 using a two group t-test with a 0.050 two-sided significance level.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients aged > or = 18 years
* Ability and willingness to adhere to the study protocol
* Signed informed consent
* Self-reported recently emerged symptoms of common cold: answer "Yes" to the question "Do you believe that you are coming down with a cold?"
* At least one of the following 4 common cold symptoms: sneezing, runny nose, nasal obstruction and/or sore throat, with no limitations of symptom severity.

Exclusion Criteria:

* Specific chronic diseases (autoimmune disease, chronic bronchitis, human immunodeficiency virus (HIV) infection, lupus, rheumatoid arthritis)
* Malignancy for which the patient has undergone resection, radiation or chemotherapy within the last five years. Patients with treated basal cell carcinoma are allowed.
* Cancer therapy
* Immunosuppressant therapies
* Use of systemic corticosteroids
* A history of asthma or allergic rhinitis and corresponding symptoms (itchy eyes, sneezing, wheezing)
* Any of the common cold symptoms persisting since more than 36 hours
* Use of other homeopathic drugs designed to treat URTIs
* Use of antibiotics, anti-histaminergic drugs or decongestants
* Participation in another clinical trial within one month prior to treatment start
* Previous participation (receipt of randomised treatment) in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Severity of symptoms of common cold | Since start of symptoms of common cold up to the visit 3 (day 10-14)
  Decrease in severity is assessed as reduction in average area under the curve (AUC) under the time severity curve (sum of all WURSS scores over the follow-up). The Wisconsin Upper Respiratory Symptom Survey-21 (WURSS-21) is a validated tool to evaluate the duration and severity of common cold. It is constituted of twenty-one categorical questions (Likert-type 7-level severity scale).

SECONDARY OUTCOMES:
Duration of common cold | Since start of symptoms of common cold up to visit 3 (Day 10-14)
  Duration is defined as the number of days from self-reported onset of disease to the last day before the participant answered "Not sick" to the question, "How sick do you feel today?" (WURSS-21). A 2-day reduction in average disease duration versus placebo will be regarded as clinically significant.
Functional impairments in the course of the disease | Since start of symptoms of common cold up to visit 3 (Day 10-14)
  Day-to-day scores for functional impairments domain. Overall (sum of all WURSS scores related to functional impairments over the follow-up).
The need of symptomatic analgesics/antipyretics | Since start of symptoms of common cold up to visit 3 (Day 10-14)
  Patients will fill in diary cards on a daily basis. The following information will be recorded: study and patient identification, date of assessment, study medication intake, other medications (name, dose, frequency) and, AEs/SAEs (description)
Evaluation of safety | since start of symptoms of common cold up to visit 3 (Day 10-14)
  Patients will fill in diary cards on a daily basis including AEs/SAEs reporting. Investigators will question patients at phone call and scheduled visits about AEs/SAEs. Frequency, severity, outcome and relationship to the study drug will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Heijmans, MD, Principal Investigator — RESEARCHLINK sprl; Luc Moriau, PhD, Study Director — ECSOR sa/nv; Michel Thiry, PhD, Study Chair — THERANOR sprl
Locations (33):
- Belgium (33):
  - Frank Heyvaert, Deurne, Antwerpen
  - Christel Van Der Geer, Geel, Antwerpen
  - Hugo Loos, Geel, Antwerpen
  - Jan Joris, Mol, Antwerpen
  - Jan De Jongh, Vorst, Antwerpen
  - Jean-Pierre Devaux, Baisy-Thy, Brabant
  - Virginie Risse, Brussels, Brabant
  - Roel De Ryck, Kraainem, Brabant
  - ResearchLink sprl, Linkebeek, Brabant
  - Stéphane Vanden Bemden, Melsbroek, Brabant
  - Bart Van Essche, Steenokkerzeel, Brabant
  - Erik Schreurs, Tremelo, Brabant
  - Lode Vermeersch, Tremelo, Brabant
  - Luc De Munck, Vilvoorde, Brabant
  - Patrice Lechien, Braine-le-Comte, Hainaut
  - Charles Corbisier, Ecaussinnes, Hainaut
  - Elise De Meulemeester, Gozée, Hainaut
  - Magali Trefois, Gozée, Hainaut
  - Aubry Robert, Ham-sur-Heure-Nalinnes, Hainaut
  - Philippe Jacques, Ham-sur-Heure-Nalinnes, Hainaut
  - Michel Grégoire, Pont-à-Celles, Hainaut
  - Etienne Demanet, Thuin, Hainaut
  - Maria Buscemi, Thuin, Hainaut
  - Etienne Plees, Beringen, Limburg
  - Nicole Olaerts, Ham, Limburg
  - Paul Beke, Leopoldsburg, Limburg
  - Steven Windmolders, Overpelt, Limburg
  - Jan Behets, Paal, Limburg
  - Jos Weckx, Paal, Limburg
  - Herman Van Den Broeck, Tessenderlo, Limburg
  - Yvan Calozet, Gribomont, Luxembourg
  - Pierre-Henri Arnould, Libramont-Chevigny, Luxembourg
  - Guy Van Damme, Heusden, Oost Vlaanderen